CLINICAL TRIAL: NCT03492723
Title: Placebo-Control, Randomized, Double Blind Long Term Trial to Evaluate the Efficacy of Garlic Product on Periodontitis
Brief Title: Garlic Product Impact on Periodontitis (GPIP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0114-17-HMO-CTIL
Record Dates: First submitted 2018-03-29; First posted 2018-04-10 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Periodontitis, Adult
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, examiner-blind, 2-treatment parallel group study.
Who Masked: Participant, Investigator
Masking Description: both, the participants and the investigators will be blind 2 groups will be assigned randomally
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- garlic groupe (Experimental): Concentrated Aged Garlic Extract Microcrystalline Cellulose 133 mg Carboxymethylcellulose Calcium 6 mg Agar Powder 35 mg Silicon Dioxide 3.5 mg Calcium Stearate 3.5 mg Total Weight 307 mg
  Interventions: Dietary Supplement: Aged Garlic Extract
- placebo groupe (Placebo Comparator): Microcrystalline Cellulose 258.55 mg Carboxymethylcellulose Calcium 6 mg Agar Powder 35 mg Coloring Agent 0.45 mg Details: Gardenia Extractive 44.5%, Corn Syrup 55% Potassium pyrophosphate 0.5% Silicon Dioxide 3.5 mg Calcium Stearate 3.5 mg Total Weight 307 mg
  Interventions: Dietary Supplement: Aged Garlic Extract

INTERVENTIONS:
Dietary Supplement: Aged Garlic Extract — NR

SUMMARY:
This is a randomized, controlled, examiner-blind, 2-treatment parallel group study. The study will be conducted at the Hebrew University, Hadassah, Israel. A sufficient number of subjects will be screened to obtain approximately 200 generally healthy adult volunteers with mild to moderate periodontitis.

Subjects will be stratified and randomly assigned equally to either the regimen group (AGE) or a control group (Placebo).

Subjects will be requested to use the products at home for the duration of the study according to the written and verbal usage instructions given to them during product distribution. At Baseline, Month 6, 12, and 18 subjects will receive oral soft tissue exams, and will have gingival inflammation, bleeding, and periodontal measurements made as described in below.

Both groups will receive supragingival dental prophylaxes every 6 month consistent with local norms and standards. Products will be re-supplied approximately every six months following Baseline. During study conduct, subjects with evidence of progressive periodontal disease (≥3 mm increases in pocket depth, attachment loss or recession) will be exited from the study and treated following local norms.

DETAILED DESCRIPTION:
Study Objective The objective of this study is to assess the long-term efficacy of "AGE among on periodontitis for a period of 2 years.

Overall Study Design and Plan This is a randomized, controlled, examiner-blind, 2-treatment parallel group study. The study will be conducted at the Hebrew University, Hadassah, Israel. A sufficient number of subjects will be screened to obtain approximately 200 generally healthy adult volunteers with mild to moderate periodontitis.

Subjects will be stratified and randomly assigned equally to either the regimen group (AGE) or a control group (Placebo).

Subjects will be requested to use the products at home for the duration of the study according to the written and verbal usage instructions given to them during product distribution. At Baseline, Month 6, 12, and 18 subjects will receive oral soft tissue exams, and will have gingival inflammation, bleeding, and periodontal measurements made as described in below.

Both groups will receive supragingival dental prophylaxes every 6 month consistent with local norms and standards. Products will be re-supplied approximately every six months following Baseline. During study conduct, subjects with evidence of progressive periodontal disease will be exited from the study and treated following local norms.

Screening/Baseline, Visit 1 Subjects will be asked to read and sign an informed consent and receive a signed copy. Personal medical history information will be reviewed and retained as site source documentation. A comprehensive oral examination (OST) will then be conducted to evaluate the oral and perioral region, including hard and soft tissues. Demographic information and study inclusion/exclusion criteria will be obtained and documented on the appropriate electronic case report form (CRF).

Then, subjects will receive MGI, GBI, CAL, and PPD assessments in that order by the experienced examiner. Subjects will be eligible to enroll in the study after meeting study entrance criteria.

Subjects will be instructed to continue using their regular home oral hygiene products until the Baseline visit. They will also be instructed not to add or change any of their regular home oral hygiene products during that time. Data will be reviewed and qualified subjects will be contacted and scheduled for their Baseline appointment. Those subjects will be asked to refrain from performing any oral hygiene procedures the morning prior to their scheduled Baseline visit and to refrain from using medicated lozenges, breath mints, eating, drinking (except for water), smoking and chewing gum for four (4) hours prior to their visit. The rest of the subjects will be released from the study, and a subject accountability form will be completed.

General Comments, if applicable, will be documented on the appropriate CRF. Product Distribution, Visit 2 Approximately maximum 1-2 weeks after the Screening/Baseline visit, subjects will return to the site and continuance criteria will be verified. Subjects will be randomized to a treatment group based on their Screening mean PPD, GBI, age, gender and tobacco use. Subjects will receive their assigned treatment products to use until their next appointment in the clinic (approximately 6 month later). AEs and General Comments, if applicable, will be documented. All data will be recorded electronically on the appropriate CRFs.

Approximately one week later, site staff not blinded to the products will re-connect to subjects via phone to ensure proper product usage and compliance.

Within one month from Baseline, subjects will receive a dental prophylaxis. Month-6, 12 Visit 3-4 Approximately 2 weeks before their scheduled visit, subjects will be contacted and reminded about their appointment. Subjects will also be reminded to bring their study products and to refrain from performing any oral hygiene procedures the morning prior to their next scheduled visit. In addition, they will be reminded to refrain from using medicated lozenges, breath mints, eating, drinking (except for water), smoking and chewing gum for four (4) hours prior to their next visit.

Subjects will return to the site (6 month from Baseline) and continuance criteria will be verified. Personal medical history information will be updated and retained as site source documentation.

A comprehensive oral examination will then be conducted to evaluate the oral and perioral region, including hard and soft tissues. Subjects will receive a MGI, GBI, CAL, and PPD assessment by the experienced examiner.

Following that, subjects will proceed to an area separated from the examination area to ensure blinding of the examiner to the identity of the test products and receive their supplemental kit box containing re-supply of their assigned treatment products. They will be asked to continue to use them for their daily oral hygiene twice per day until their next appointment in the clinic (approximately 6 month later). Instructions for home use and a reminder to comply with the study protocol will be given verbally by the site staff.

AEs and General Comments, if applicable, will be documented. All data will be recorded electronically on the appropriate CRFs.

Within one month from Month-6 visit, subjects will receive a dental prophylaxis.

Month-18, Visit 5 Approximately 2 weeks before their scheduled visit, subjects will be contacted and reminded about their appointment. Subjects will also be reminded to bring their study products and to refrain from performing any oral hygiene procedures the morning prior to their next scheduled visit. In addition, they will be reminded to refrain from using medicated lozenges, breath mints, eating, drinking (except for water), smoking and chewing gum for four (4) hours prior to their next visit.

Subjects will return to the site (18 month from Baseline) and continuance criteria will be verified. Personal medical history information will be updated and retained as site source documentation.

A comprehensive oral examination will then be conducted to evaluate the oral and perioral region, including hard and soft tissues. Subjects will receive a MGI, GBI, CAL, and PPD assessment by the experienced examiner.

AEs and General Comments, if applicable, will be documented. Subject accountability will be completed and subjects will be dismissed from the study. Subject accountability will also be completed for subjects who drop out of the study prior to its completion.

All data will be recorded electronically on the appropriate CRFs.

ELIGIBILITY:
Inclusion Criteria

* give written informed consent and receive a copy of their consent
* be between the ages of 30 to 60 years
* be in good general health as determined by the Investigator or designee
* based on a review of the medical history or update for participation in the study
* possess a minimum of 16 natural teeth with facial and lingual scorable surfaces
* have at least 20 bleeding sites
* have at least 3 eligible periodontal sites
* agree to delay any elective dentistry until study completion, including additional dental prophylaxes outside the study protocol
* agree to refrain from using any non study oral hygiene products for the study duration
* agree not to participate in any other oral care clinical study for the duration of this study
* agree to return for their scheduled visits and follow study procedures

Exclusion Criteria

* severe periodontal disease, as characterized by purulent exudate, generalized mobility, and or severe recession
* active treatment for periodontitis
* having a medical condition requiring antibiotic premedication prior to dental procedures,
* fixed facial or lingual orthodontic appliances or removable partial dentures
* antibiotic or chlorhexidine use or antiinflammatory medications within two weeks prior to Screening visit
* self report nursing, pregnancy, or intent to become pregnant during the study
* dental prophylaxis within two month prior to the Screening visit
* any diseases or conditions that could be expected to interfere with the subject safely completing the study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-04-17 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevention of Gindivitis | 4 months
  A reduction of bleeding index in the Garlic group
Prevention of Gindivitis | 4 months
  A reduction of Gingival index in the Garlic group

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Mann, DMD, Principal Investigator — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Hadassah Medical Organization,, Jerusalem
  - Hadassah Medical Organization, Jerusalem

IPD SHARING:
Plan to Share IPD: No
the data will not be available to other researcher and will be save under personal password